CLINICAL TRIAL: NCT00921427
Title: The Use of Transcranial Direct Current Stimulation (TDCS) to Enhance the Rehabilitative Effect of Vision Restoration Therapy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Lotfi Merabet, PI, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007-P-000241
Record Dates: First submitted 2009-06-14; First posted 2009-06-16 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Hemianopia; Quadrantanopia; Scotoma; Visual Field Loss
Keywords: Hemianopia; Rehabilitation; Transcranial direct current stimulation; Visual field
MeSH Terms: conditions — Hemianopsia; Scotoma | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VRT and active tDCS (Active Comparator): Patients will receive tDCS (noninvasive brain stimulation) concurrently with vision restoration therapy. TDCS is delivered using a small battery-operated device. Electrical leads from the device are connected to saline soaked sponges that are placed at strategic locations on the skull corresponding to areas of the brain that need to be stimulated (in this case, the visual cortex). The dosage will be set to 2 mA/min for 30 minutes, twice a day for 3 days a week for 12 weeks.
  Interventions: Behavioral: Vision Restoration Therapy (VRT); Device: Transcranial direct current stimulation (tDCS)
- VRT combined with sham tDCS (Sham Comparator): Patients will receive sham tDCS concurrently with vision restoration therapy. Electrical leads from the tDCS device will be connected to saline soaked sponges placed at strategic locations on the skull, in a similar maner as in the active tDCS group. Current will be turned on for 30 seconds but will be slowly ramped down and turned off. Treatment will continue for 3 days a week for 12 weeks.
  Interventions: Behavioral: Vision Restoration Therapy (VRT)

INTERVENTIONS:
Behavioral: Vision Restoration Therapy (VRT) — 30 min, twice a day, 3 days a week, 12 weeks
Device: Transcranial direct current stimulation (tDCS) — 2 mA/min, 30 min, twice a day, 3 days a week for 12 weeks
  Arms: VRT and active tDCS

SUMMARY:
The purpose of our study is to explore the efficacy of combination of brain stimulation with visual rehabilitation in patients with visual field loss resulting from brain lesions. It is shown that the effect of sensorimotor training of hand can be enhanced in patients with stroke using brain stimulation. We decided to explore this combination for visual field loss because visual dysfunction following brain lesions is considered intractable. We hypothesize that combination of noninvasive brain stimulation, in the form of transcranial direct current stimulation (tDCS), with visual rehabilitation would have greater efficacy than visual rehabilitation alone.

DETAILED DESCRIPTION:
The specific aim of this study is to improve recovery of visual function after brain injury. A prominent theme of current neuroscience research regarding the sequelae of brain injury posits that activity-dependent plasticity underlies neuro-recovery. If that is the case, there is good reason to believe that neurological changes underling recovery can be facilitated by established means of enhancing cortical activity. Studies suggest that altering cortical excitability may prime or prepare the cortex for subsequent training and furthermore, may improve overall functional outcomes (Webster et al, 2006; Brown & Pilitsis, 2006; Khedr et al, 2005). The working hypothesis of this pilot study is that computer-based visual rehabilitative training (using NovaVision's Vision Restoration TherapyTM; "VRT" software) enhances visual function (defined as an increase in functional visual field) by reinforcing synaptic connections within sensory networks of visual cortex associated with the visual field loss (Kasten et al., 1998; Sabel, 1999). Potentially, this reinforcement can be enhanced by concurrent transcranial direct current stimulation (TDCS) leading in turn, to enhanced visual performance (quantified by the extent of visual field measured by visual perimetry allowing for a direct statistical comparison of visual field change over time and on an individual basis) in patients with partial of complete hemianopic visual field loss caused by brain injury. Both computer based visual rehabilitative training and TDCS are established techniques and this novel approach aims to provide preliminary data regarding the safety and efficacy of a combined intervention.

We expect that results from this study will provide an objective basis for a larger, formal randomized controlled study combining the two therapies. Our long term goals are to maximize the benefits of a modern vision rehabilitative therapy, lay the groundwork for neurophysiological correlates associated with the recovery of visual function following brain injury and propose possible refinements for future neurorehabilitation strategies. Data from our collaborators at Columbia University Medical Center as well as others indicate that a 6 month course treatment therapy of VRT can lead to dramatic improvements in visual function (as quantified by increases in functional visual field) (Kasten et al., 1998; Kasten et al., 2006). TDCS is well known to bring about transient positive changes in both functional as well as electrophysiological measures of cortical brain function. If overall visual function can be further enhanced via a combined synergetic effect of VRT and TDCS, we will conduct a larger randomized controlled study. If there is no enhancement effect with combined TDCS and VRT, we will need to reconsider factors as to why this is the case. For example, a lack of enhancement effect could be related to patient selection including the degree and profoundness of vision loss prior to treatment, the age of the individual and duration of the insult, as well as their level of motivation in participating with the computer-based training program. Other considerations include longer combined treatment duration.

The loss of visual function following brain injury can be highly debilitating for an individual. Typically, damage to the occipital cortex or optic radiations following a brain lesion or trauma leads to a loss of visual function in visuotopically corresponding parts of the visual field while sparing the remaining areas (e.g. half the visual field as in the case with hemianopia). This partial blindness and loss in visual function has generally been considered untreatable due to the fact that the highly specific neuronal organization underlying normal visual function is determined early in development and not regenerative particularly after the "critical period" of development has been reached. More recent evidence (including that from our laboratory) has demonstrated that a considerable degree of plasticity and reorganization of the visual system occurs not only after cerebral damage but also in adulthood, that is, well after the critical period of development has occurred. For example, evidence of spontaneous post-lesion neuroplasticity has been demonstrated in the adult visual system as documented by extensive receptive field reorganization following lesions in the retina or visual cortex (e.g. Kass 1990).

Computer-based training strategies have been developed to train and rehabilitate various cerebral functions such as language learning deficits. Computer-based training has also been extensively studied as a treatment for partial blindness in adult brain-injured patients (Kasten et al., 1998; Sabel and Trauzettel-Klosinksi, 2005; Sabel et al., 2005). However, the neurophysiological mechanisms underlying the reported beneficial effect following VRT remains poorly understood. One important issue is that if the restoration of visual field and function is the result of localized neuroplastic changes in cortical circuitry within visual cortex, one can posit that modulation of cortical excitability should in turn influence the degree of this restorative effect. More specifically, increasing the level of overall cortical excitability of the visual cortex should potentiate synaptic neuroplastic interactions and thus translate into improved visual functional gains.

Transcranial Direct Current Stimulation (TDCS) represents a noninvasive method of brain stimulation that could potentially modulate such an effect. TDCS utilizes low amplitude direct currents applied via scalp electrodes to inject currents in the brain and thus modulate the level of excitability. Direct Current (DC) stimulation has been used in various forms since the inception of modern electrophysiology at the beginning of nineteenth century. There has been a recent upsurge in interest in TDCS as a tool for neuroscience research as well as an assessment and treatment modality for various neurological and neuropsychiatric disorders including depression, Parkinsonism, stroke recovery, and chronic neuropathic pain. TDCS has the distinct advantage of being inexpensive, easy to administer, noninvasive and painless. We have extensive experience with TDCS and are currently running parallel studies. We now wish to extend these principles into the visual rehabilitation domain.

VRT: Computer-based training strategies have been developed to train and rehabilitate adult brain-injured patients with partial visual loss due to brain damage (Kasten et al., 1998; Sabel and Trauzettel-Klosinksi, 2005; Sabel et al., 2005). Vision restoration therapy (VRT) involves identifying and stimulating regions in the visual field that are only partly damaged by brain injury or trauma. Patients receive a customized program designed for their visual field deficits to use at home daily. Through a specific pattern of visual stimuli that gauge the user's ability to identify and react, users can gradually expand their visual fields and restore lost vision. The training can be done at home in front of a computer-based device, usually in 30-minute sessions, twice a day. During the training, hundreds of visual stimulations are presented on the monitor to the areas of residual vision. It has been proposed that repetitive stimulation of damaged visual areas leads to neuroplastic changes altering nerve activity related to vision, and strengthening synaptic interactions that can help restore some of a person's visual functions. Work by Sabel and colleagues reported findings from fifteen patients that underwent six and 12 months of VRT (Kasten et al., 2006). Visual field assessments were performed before and after VRT and then repeated an average of 46 months after completing VRT. After six months of VRT, sample stimulus detection increased significantly from about 54% to 63%. The number of undetected stimuli decreased significantly in both eyes. Continuing VRT for 12 months improved the results achieved at six months. The follow-up examination after a therapy-free interval of more than three years showed that the benefits of VRT remained stable, and vision loss did not occur in most instances. According to this study, patients with vision loss after brain injury benefit regardless of the severity of the lesion or how much of their vision is affected. Furthermore, the larger the areas of residual vision, the better the outcome with VRT. It is clear that VRT has varying results. In this study, one-third of patients studied had little or no effect from VRT, one-third had moderate but noticeable improvement, and one-third had strong or dramatic improvement. Patient compliance with VRT is reported to be very good.

NovaVision VRT™ is the first and only FDA-cleared medical device or rehabilitative therapy clinically proven to improve visual field defects in brain injury survivors who have become left partially blind due to their condition. In an on-going multi-center trial sponsored by NovaVision, over 70% of study participants from 16 U.S. centers who underwent a six-module (six month) course of therapy showed a three percent or greater improvement in stimulus detection on visual field testing. The average improvement in stimulus detection was 12 percent. Previous studies suggest that people who regain three percent or more of their visual field have functional improvements that may include enhanced quality of life through better reading performance, watching television and playing sports, although functional outcomes were not measured in this study. These results were presented at the 2007 Academy of Neurology meeting in Boston, MA.

TDCS: Transcranial direct current stimulation (TDCS) has been used for several decades. Numerous human clinical and animal studies have demonstrated that this technique is able to modulate neuronal activity and function through the delivery of polarizing currents applied to the surface of the brain. Surface anodal polarization of the cortex increases spontaneous neuronal activity, whereas cathodal polarization generally depresses neuronal activity (Creutzfeld et al., 1962). Recent human studies have demonstrated that stimulation with TDCS changes motor cortex excitability according to the stimulation polarity: whereas anodal stimulation increases cortical excitability, cathodal stimulation decreases it (Nitsche et al., 2003a and b). Moreover, and from a clinical therapeutic point of view, the effects of TDCS appear to be long-standing. For example, 13 minutes of TDCS has been shown to modulate cortical excitability and last up to 2 hours following the stimulation period itself (Nitsche and Paulus, 2001). Two recent studies (including one by a co-investigator listed here) explored the effects of TDCS on motor function in stroke patients and showed that these modulatory effects of TDCS can be used to improve motor function (Fregni et al., 2005a; Hummel et al., 2005a and b). Interestingly, similar modulatory effects have also been described in the visual cortex (Antal et al., 2001; Antal et al., 2004) leading support to the notion that activity within visual cortical areas can be modulated and in turn lead to behavioral changes.

TDCS modulates the excitability of a targeted brain region non-invasively by altering neuronal membrane potentials (Bindman et al. 1962; Purpura & McMurtry, 1965). Thus, this technique can be used to increase or decrease the excitability of neurons in a targeted brain area and this can establish a causal relation between a given region of the brain and a specific sensory, motor or cognitive function. Unlike Transcranial Magnetic Stimulation (TMS), TDCS does not depolarize neurons causing them to fire. TDCS only alters the likelihood that neurons will fire by depolarizing or hyperpolarizing brain tissue (depending on the stimulation parameters used). The neurophysiological basis of TDCS has been attributed to a mechanism akin to long-term potentiation (LTP) and long-term depression (LTD) (Hattori et al. 1990; Moriwaki, 1991; Islam et al. 1995). Certain medications such as dextromethorphan (an NMDA antagonist) suppress post-TDCS stimulation effects of both anodal and cathodal stimulation which strongly suggests the involvement of NMDA receptors in both types of DC-induced neuroplasticity. In contrast, Carbamazepine selectively eliminates anodal effects. Since Carbamazepine stabilizes the membrane potential voltage-dependently, the results reveal that after-effects of anodal TDCS require a depolarization of membrane potentials (Liebetanz et al., 2002). This study by Liebetanz et al., (2002) provided pharmacological evidence that induction of the after-effects of TDCS requires a combination of glutamatergic (excitatory) and membrane mechanisms, similar to the induction of established types of short- or long-term neuroplasticity.

In animals, anodal cortical stimulation of 5-30 minutes has been shown to cause excitability increases lasting for hours after the stimulation, primarily through modulation of the resting membrane potential (Terzuolo & Bullock, 1956; Creutzfeldt et al. 1962; Eccles et al. 1962; Bindman et al. 1964; Purpura & McMurtry, 1965; Artola et al. 1990; Malenka & Nicoll, 1999). In humans, 13 min of TDCS resulted in an increase in excitability up to 150% and lasting 90 min (Nitsche & Paulus, 2001). Research with TDCS has revealed that anodal stimulation can induce transient (on the order of 30 minutes) improvements in performance on cognitive, motor and linguistic tasks. For example, Hummel et al. (2005a,b) found that anodal TDCS delivered to the primary motor area in the lesion hemisphere elicited significant improvements in motor control of the paretic limb. The effect lasted for more than 25 minutes after stimulation. In a recent study, Fregni et al (2005a) also verified that anodal TDCS to the affected hemisphere and cathodal TDCS to the contralesional hemisphere improved motor function. Other examples highlighting the efficacy of anodal TDCS include Fregni et al. (2005b) - anodal TDCS to dorsolateral prefrontal cortex elicited an improvement in working memory; Nitsche et al. (2003a) - stimulation to primary motor cortex improved motor learning; Antal et al. (2004) - TDCS delivered to primary motor area or to visual area V5 induced improvements in visuo-motor coordination; Kincses et al. (2004) - anodal stimulation of fronto-polar regions improved probabilistic classification learning; and Lyer et al. (2005) - left prefrontal cortical stimulation lead to increased verbal fluency. These studies attest to the efficacy and safety of TDCS in brain injury patients, as well as its potential for therapeutic applications in brain lesion recovery.

In summary, we propose to conduct a pilot experiment testing whether visual function in-patients with hemianopic field loss caused by brain injury can be improved by combining transcranial direct stimulation and computer based vision training. We hypothesize that computer based vision training will reinforce visual cortical networks primed by concurrent transcranial direct current stimulation (TDCS) and lead to improved visual performance. The BIDMC investigators will be responsible for TDCS application and VRT, as well as associated data processing / interpretation.

ELIGIBILITY:
Inclusion Criteria:

* Hemianopic field loss is defined as (a) visual field defect on the same side of visual space in both eyes as determined by monocular perimetry and (b) established structural damage of the post-charismatic visual system as documented by standard neuroimaging techniques (CT or MRI), medical reports, or a combination of these
* deep scotoma - defined field loss as confirmed by perimetry
* cognitive, language and motor function sufficient to understand the experiments and follow instructions
* informed written consent to participate in the study
* motivation to participate in the VRT program

Exclusion Criteria:

* any sensory-motor loss other than visual
* ongoing use of CNS-active medications for an active neurological disease
* ongoing use of psychoactive medications, such as stimulants, antidepressants, and anti-psychotic medications for an active psychiatric condition
* presence of additional potential TDCS risk factors:

  * Damaged skin at the site of stimulation (i.e., skin with ingrown hairs, acne, razor nicks, wounds that have not healed, recent scar tissue, broken skin, etc.)
  * Presence of an electrically, magnetically or mechanically activated implant (including cardiac pacemaker), an intracerebral vascular clip, or any other electrically sensitive support system.
  * Metal in any part of the body, including metal injury to the eye. (Jewelry must be removed during stimulation.)
  * A history of medication-resistant epilepsy in the family
  * Past history of seizures or unexplained spells of loss of consciousness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-11; Primary Completion 2010-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Visual Field Gain in Degrees | Once every month for three months

SECONDARY OUTCOMES:
Visual Field test- Percent accuracy of detection | Once every month for three months
Functional Questionnaire (Impact of Vision Impairment Profile) | Once every month for three months
Subjective Drawing of the Visual Field (area of blind field in sq. mm) | Once every month for three months

CONTACTS AND LOCATIONS:
Overall Officials: Lotfi B Merabet, OD PhD, Principal Investigator — Beth Israel, Harvard Medical School; Alvaro Pascual-Leone, MD PhD, Study Director — Beth Israel, Harvard Medical School, Neurology